CLINICAL TRIAL: NCT01245946
Title: Efficacy Comparison Study of Topical Aminolaevulinic Acid-Photodynamic Therapy Versus Adapalene Gel 0.1% Plus Doxycycline for Treatment of Moderate Acne Vulgaris. Randomized, Simple Blind, Controlled Trial.
Brief Title: Photodynamic Therapy Compared to Adapalene 0.1% Gel Plus Doxycycline in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Claudia Nicklas D, Department of Dermatology, Pontificia Universidad Católica de Chile, Pontificia Universidad Católica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-146
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2010-11

CONDITIONS: Acne
Keywords: Acne moderate; Photodynamic Therapy; Topical retinoids; Antimicrobial agents
MeSH Terms: conditions — Acne Vulgaris | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Adapalene; Doxycycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Photodynamic therapy (Experimental)
  Interventions: Procedure: Photodynamic therapy
- Conventional therapy (Experimental)
  Interventions: Drug: Conventional therapy

INTERVENTIONS:
Procedure: Photodynamic therapy — Photodynamic therapy: 2 sessions separated by 2 weeks of TDF with topical ALA20% for 1.5 hrs, then irradiated with red light (Waldmann lamp) at a fluence of 37 J/cm2 for 7-9 minutes. From the sixth week will begin adapalene 0.1% gel until 12 weeks
  Other Names: PDT
  Arms: Photodynamic therapy
Drug: Conventional therapy — Conventional therapy: Topical adapalene gel 0.1% at night for 12 weeks plus doxycycline 100 mg / day for 6 weeks.
  Other Names: Adapalene plus doxycycline
  Arms: Conventional therapy

SUMMARY:
* Acne vulgaris is a common inflammatory skin disease that affects more than 85% of teens and some people may continue throughout adulthood.
* Topical retinoids related to oral antibiotics are considered first-line treatment of moderate inflammatory acne.
* Recently, photodynamic therapy (PDT) with a photosensitizer, 5-aminolevulinic acid (ALA) or methyl aminolevulinate (MAL), has proven useful in the management of inflammatory acne. Although progress has been made in the study of photodynamic therapy for acne, to date, no study has compared PDT with standard and well-validated pharmaceutical treatments and with the current recommended therapy for most types of acne combination therapy with a topical retinoid plus one or more antimicrobial agents.

Hypothesis

* PDT with the photosensitizer ALA will be effective and safe for the treatment of moderate facial inflammatory acne.
* The ALA-PDT is more effective than conventional therapy with oral antibiotics and topical retinoids in the treatment of moderate inflammatory acne with faster action at 12 weeks of follow-up.

DETAILED DESCRIPTION:
* There will be a randomized, controlled, single blind comparison study of PDT with 5-aminolevulinic acid (ALA) 20% versus conventional therapy consisting of topical 0.1% adapalene plus doxycycline 100 mg/day orally in patients with moderate inflammatory acne.
* Be sought from all patients written informed consent prior to study entry.
* For sample size calculation, we assumed that the correlation is the same in both groups and is relatively low (0.01), the number of lesions per subject is equal in both groups with a mean of 100 and low variance, which take 1 control per case and that. Whereas the percentage of improvement in the control group is 0.6 and expected in the treatment group is 0.7 yields a sample size of 23 patients in the treatment group and 23 new controls.

Interventions:

Patients will be randomized to receive:

1. ALA-PDT: In 23 patients applied 20% ALA solution in the affected area for 1.5 hours. Subsequently irradiated with noncoherent red light (lamp Waldmann PDT 1200; wavelength 590-700 nm) with irradiance of 70 mW/cm2 and total dose or fluence of 37 J/cm2 for 7-9 minutes. From the sixth week will begin nightly topical adapalene 0.1% gel.
2. Standard therapy:

In 23 patients applied topical adapalene 0.1% gel at night for 12 weeks plus doxycycline 100 mg / day for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 30 years of age with moderate inflammatory acne

Exclusion Criteria:

* Those who have received any treatment for acne either topic in the last 3 months before and systemic (including ACO started) in the last 6 months of the study.
* Patients who are pregnant or breastfeeding.
* Patients with history of photosensitivity or autoimmune disease.
* Patients with a history or active TB disease or HIV.
* Patient refusal to participate in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Lesion counts | Twelve weeks
  Be conducted by an investigator blinded to the interventions, count of inflammatory and non-inflammatory acne lesions at the start of treatment and controls at the sixth and twelfth week.

SECONDARY OUTCOMES:
Photographic scores, quality of life, adherence to treatment and global severity of acne | Twelve weeks
  The researchers will make assessment of the quality of life, adherence to treatment, global severity of acne and scars and blemishes record at the beginning and end of the study (12 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Hasson, MD, Study Chair — Dermatology department, Pontificia Universidad Católica de Chile
Locations (1):
- Departamento de dermatología, Centro Médico San Joaquín, Pontificia Universidad Católica de Chile, Santiago, San Joaquín, Chile